CLINICAL TRIAL: NCT05994599
Title: SINGLE DOSE CROSSOVER COMPARATIVE BIOAVAILABILITY STUDY OF ETHINYL ESTRADIOL/ETONOGESTREL VAGINAL RING (DELIVERING 0.015 mg/0.12 mg PER DAY) WORN FOR 21 DAYS IN HEALTHY FEMALE SUBJECTS
Brief Title: Comparative Bioavailability Study of Ethinyl Estradiol/Etonogestrel Vaginal Ring
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evestra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: EVE-P6-604
Record Dates: First submitted 2023-08-01; First posted 2023-08-16 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Healthy Women; Female; Contraception

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Laboratory Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- EVE119 vaginal ring (Experimental): EVE119 (ethinyl estradiol/etonogestrel) vaginal ring delivering 0.015 mg/0.12 mg dose per day
  Interventions: Combination Product: EVE119 vaginal ring
- Nuvaring vaginal ring (Active Comparator): Nuvaring® (ethinyl estradiol/etonogestrel) vaginal ring delivering 0.015 mg/0.12 mg dose per day
  Interventions: Combination Product: Nuvaring vaginal ring

INTERVENTIONS:
Combination Product: EVE119 vaginal ring — EVE119 (ethinyl estradiol/etonogestrel) vaginal ring delivering 0.015 mg/0.12 mg dose per day
  Arms: EVE119 vaginal ring
Combination Product: Nuvaring vaginal ring — Nuvaring® (ethinyl estradiol/etonogestrel) vaginal ring delivering 0.015 mg/0.12 mg dose per day
  Arms: Nuvaring vaginal ring

SUMMARY:
Single Dose Crossover Comparative Bioavailability Study of Ethinyl Estradiol/Etonogestrel Vaginal Ring (Delivering 0.015 mg/0.12 mg Per Day) Worn for 21 Days in Healthy Female Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated Informed Consent Form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Healthy adult female
4. Meets 1 of the following criteria:

   1. Is of childbearing potential and agrees to use an acceptable contraceptive method. Acceptable contraceptive methods include:

      * Abstinence from heterosexual intercourse from the Screening visit through to at least 28 days after the last vaginal ring removal
      * The following double-barrier contraceptive methods, used from the Screening visit through to at least 28 days after the last vaginal ring removal:

        * Male condom with spermicide Or
   2. Is of non-childbearing potential, defined as surgically sterile (ie, tubal ligation)
5. Aged at least 18 years but not older than 45 years in pre-menopausal state
6. Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively
7. Non- or ex-smoker (An ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first vaginal ring insertion)
8. Normal pap test result on file at Altasciences in the previous 12 months prior to the first vaginal ring insertion or normal pap test result at Screening
9. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including breast and gynecological examination) and/or electrocardiogram (ECG), as determined by an Investigator

Exclusion Criteria:

1. Female who is lactating
2. Female who is pregnant according to the pregnancy test at Screening or prior to the first vaginal ring insertion
3. Use of the following systemic contraceptives: oral, patch, or vaginal ring, in the 28 days prior to the first vaginal insertion and until completion of the study
4. Use of hormone replacement therapy in the 28 days prior to the first vaginal insertion and until completion of the study
5. Use of the following systemic contraceptives: injections or implant, or hormone-releasing intrauterine device (IUD) in the 13 weeks prior to the first vaginal insertion and until completion of the study
6. Has contraindication for contraceptive steroids
7. Post-menopausal status (minimum of a year without menses) and/or has undergone a complete hysterectomy or bilateral oophorectomy
8. Seated blood pressure higher than 140/90 mmHg at the Screening visit and prior to the first vaginal ring insertion, unless deemed non-significant by an Investigator
9. History of significant hypersensitivity to ethinyl estradiol, etonogestrel, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
10. Presence or history of significant genital, gastrointestinal, liver or kidney disease, or any other condition that is known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
11. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease, as defined by the Investigator
12. Presence of clinically significant ECG abnormalities at the Screening visit, as defined by the Investigator
13. Known presence or history of thrombophlebitis or any thromboembolic disorders (eg, venous thrombosis, arterial thrombosis), with or without pulmonary embolism
14. Known predisposition for venous or arterial thrombosis, with or without hereditary involvement such as Activated Protein C-resistance (including Factor V Leiden), antithrombin-III deficiency, protein C deficiency, protein S deficiency, hyperhomocysteinemia, and antiphospholipid antibodies (anticardiolipin antibodies, lupus anticoagulant)
15. Known presence or history of classic migraine
16. Known presence of ocular lesion arising from ophthalmic vascular disease, such as partial or complete loss of vision or defect in visual fields
17. Known presence, suspected presence or history of cervical, breast, uterine, estrogen-dependent, or progestin-dependent cancer or other sex-steroid sensitive malignancies
18. Known presence or history of undiagnosed abnormal vaginal bleeding
19. Known presence of any condition that makes the use of the vaginal ring difficult such as prolapse of the uterine cervix, cystocele, and/or rectocele, severe or chronic constipation
20. Any other vaginal condition that would interfere with the vaginal ring or cause an increased health risk
21. Scheduled immunization with a Coronavirus Disease 2019 (COVID-19) vaccine during the study that, in the opinion of an Investigator, could potentially interfere with subject participation, subject safety, study results, or any other reason
22. Major surgery with prolonged immobilisation in the previous 6 months prior to the first vaginal ring insertion
23. Planned major elective surgery in the 3 months following removal of the vaginal ring
24. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
25. Any clinically significant illness in the 28 days prior to the first vaginal ring insertion
26. Use of any prescription drugs in the 28 days prior to the first vaginal ring insertion, that in the opinion of an Investigator would put into question the status of the participant as healthy
27. Use of St. John's wort in the 28 days prior to the first vaginal ring insertion
28. Any history of tuberculosis
29. Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first vaginal ring insertion
30. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen, or hepatitis C virus tests
31. Serum ferritin value below 24 μg/L at Screening
32. Any other clinically significant abnormalities in laboratory test results at Screening that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
33. Inclusion in a previous group for this clinical study
34. Intake of ethinyl estradiol or etonogestrel in the 28 days prior to the first vaginal ring insertion
35. Intake of an IP in the 28 days prior to the first vaginal ring insertion
36. Donation of 50 mL or more of blood in the 28 days prior to the first vaginal ring insertion
37. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first vaginal ring insertion
38. Hemoglobin laboratory values below the lower limit of the reference at Screening -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2023-07-29 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence: evaluate and compare the bioavailability and therefore to assess the bioequivalence of 2 different formulations of ethinyl estradiol/etonogestrel vaginal ring | Up to 24 days post ring insertion per period
  The primary study endpoints are the pharmacokinetic (PK) parameter is the Cmax.
Bioequivalence: evaluate and compare the bioavailability and therefore to assess the bioequivalence of 2 different formulations of ethinyl estradiol/etonogestrel vaginal ring | Up to 24 days post ring insertion per period
  The primary study endpoints are the pharmacokinetic (PK) parameter is AUC0-T of ethinyl estradiol and etonogestrel.
Bioequivalence: evaluate and compare the bioavailability and therefore to assess the bioequivalence of 2 different formulations of ethinyl estradiol/etonogestrel vaginal ring | Up to 24 days post ring insertion per period
  The primary study endpoints are the pharmacokinetic (PK) parameter is and AUC0-∞ of ethinyl estradiol and etonogestrel.

SECONDARY OUTCOMES:
Safety and tolerability of the vaginal rings | through study completion, expected 102 days
  Incidence and severity of treatment emergent adverse events (TEAEs) and serious TEAEs
Evaluate the vaginal local irritation and occurrence of bleeding/spotting | through study completion, expected 102 days
  Assessment of vaginal irritation and occurrence of bleeding/spotting through subject questionnaire/diary.

CONTACTS AND LOCATIONS:
Overall Officials: Ze'ev Shaked, PhD, Study Director — Evestra CEO
Locations (1):
- Altasciences, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No